CLINICAL TRIAL: NCT03684226
Title: Stroke Observatory of Caen-Normandie Metropole
Acronym: NORMANDYSTROKE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 17-007
Record Dates: First submitted 2018-06-07; First posted 2018-09-25 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2018-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stroke Observatory of Caen-Normandy Metropole provides epidemiological data in prospective collection. The primary objective is to determinate incidence of Stroke in this area. Several data sources will be crossed to allow an exhaustive identification of the cases. No intervention will be carried. The data collected will correspond to those obtained in current practice. The number of participants is estimated at 800 per year. This Observatory aims to become a qualified population register after three years, according to requirement of the french registry evaluation committee.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death (the first in women in industrialized countries), the second cause of dementia and the third leading cause of disability. For a middle-aged person, the risk of developing a stroke is 1/5 in women and 1/6 in men over a lifetime. Moreover, stroke is a disease that can be considered chronic. Indeed, in France, the survival rate one month after a stroke is 80-90%. However, at least 50% of survivors retain a severe disability and almost all require long-term care. The medico-economic impact of stroke is therefore important in both the initial and chronic phases. Nevertheless, none of the French stroke registries consider the burden of post-stroke disability. In addition, there is limited data available on the impact of geographic disparities on the prognosis of stroke. Population studies are essential to accurately identify the incidence and burden of stroke, thereby supporting public health policy, guiding the allocation of resources, and evaluating the effectiveness of preventive strategies for a population. This is why we propose to create a Norman Observatory of Stroke. It will include an urban and rural population and will aim to become a population register.

ELIGIBILITY:
Inclusion Criteria:

* Any types of strokes (initial, recidivism)
* Place of residence in Caen-Normandie Metropole
* Age higher than 30 days (exclusion of perinatal stroke)

Exclusion Criteria:

* None, unless patient opposition

Min Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Caen-Normandie Metropole is a territory that includes one hundred forty five municipalities with urban, peri-urban and rural area. Total population is approaching 800 000 inhabitants
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2017-05-17 (Actual); Primary Completion 2020-05-17 (Estimated); Study Completion 2020-05-17 (Estimated)

PRIMARY OUTCOMES:
Stroke incidence in Caen-Normandy Metropole | 15 may 2017 to 15 may 2020
  To determinate the incidence of stroke in Caen-Normandy Metropole
Stroke acute mortality in Caen-Normandy Metropole | 15 may 2017 to 15 may 2020
  To determinate the incidence of Stroke acute mortality

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel TOUZE, MD, Principal Investigator — CHU of CAEN
Locations (1):
- CHU of CAEN, Caen, France

IPD SHARING:
Plan to Share IPD: No